CLINICAL TRIAL: NCT01561846
Title: Randomized, Double Blind, Controlled, Cross Over Clinical Trial on Intake of CLA Enriched Cheese in Hypercholesterolemic Patients
Brief Title: Cheese Intake,CLA and Hypercholesterolemia
Acronym: CASU
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliera Brotzu (Other)
Collaborators: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Pintus, Medical Doctor, Azienda Ospedaliera Brotzu
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AOBROTZUCMDA
Record Dates: First submitted 2012-03-22; First posted 2012-03-23 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Modifications of LDL Cholesterol; Modifications of Enocannabinoid Levels
Keywords: Conjugated Linoleic Acid; LDL-cholesterol; Endocannabinoids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- regular cheese (Active Comparator): This study was a 3-week, randomized, double blind, controlled, cross over clinical trialy. The subjects were randomly assigned to eat 90g/d of the control or enriched cheese for 3 weeks, with a cross over after 3 weeks of washout. The study included 5 visits: 2 screening/baseline visits at weeks -1 and 0, 1 end of intake of 90 g/d of cheese visit at week 3, 1 end of the first wash out visit at week 6, and 1 end of treatment after crossing over visit at week 9. This procedure was subsequently repeated with a cheese intake of 45 g/d
  Interventions: Dietary Supplement: CLA enriched cheese
- CLA enriched cheese (Experimental)
  Interventions: Dietary Supplement: CLA enriched cheese

INTERVENTIONS:
Dietary Supplement: CLA enriched cheese — This study was a 3-week, randomized, double blind, controlled, cross over clinical trial, conducted at the State Hospital Brotzu in Cagliari, Italy. The subjects were randomly assigned to eat 90g/d of the control or enriched cheese for 3 weeks, with a cross over after 3 weeks of washout. The study included 5 visits: 2 screening/baseline visits at weeks -1 and 0, 1 end of intake of 90 g/d of cheese visit at week 3, 1 end of the first wash out visit at week 6, and 1 end of treatment after crossing over visit at week 9. This procedure was subsequently repeated with a cheese intake of 45 g/d
  Arms: regular cheese
Dietary Supplement: CLA enriched cheese — This study was a 3-week, randomized, double blind, controlled, cross over clinical trial, conducted at the State Hospital Brotzu in Cagliari, Italy. The subjects were randomly assigned to eat 90g/d of the control or enriched cheese for 3 weeks, with a cross over after 3 weeks of washout. The study included 5 visits: 2 screening/baseline visits at weeks -1 and 0, 1 end of intake of 90 g/d of cheese visit at week 3, 1 end of the first wash out visit at week 6, and 1 end of treatment after crossing over visit at week 9. This procedure was subsequently repeated with a cheese intake of 45 g/d

SUMMARY:
In this study the investigators aimed at verifying whether consumption of a sheep cheese, naturally enriched in ALA, CLA and VA, would modify the plasma lipid and endocannabinoid profiles in mild hypercholesterolemic subjects. This study was a 3-week, randomized, double blind, controlled, cross over clinical trial, conducted at the State Hospital Brotzu in Cagliari, Italy. The subjects were randomly assigned to eat 90g/d of the control or enriched cheese for 3 weeks, with a cross over after 3 weeks of washout.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers with diagnosed mild hypercholesterolemia (total cholesterol 220-290 mg/dL)

Exclusion Criteria:

* Pregnant (or those planning to become pregnant during the study period) and lactating women
* Also individuals with a self-reported history of diabetes, inflammatory bowel disease, pancreatitis, gallbladder or biliary disease in the past 12 months, and lactose intolerance before the screening visit.
* Those with a history of cancer (except non-melanoma skin cancer) in the 2 years before screening, or of any major trauma or surgical event within 3 months before screening.
* Volunteers with the following characteristics were also excluded:

  * total cholesterol ≥300 mg/dL, serum triglycerides ≥250 mg/dL or ≤ 200 mg/dL, *HDL ≥70mg/dL, BMI ≥ 30
  * uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) at screening.
* Use of lipid-altering medications or supplements, and of anticoagulants, during the 2 weeks before screening and throughout the study was prohibited.
* Furthermore, we selected subjects with an Apo E aplotype 3/3, the most common in Sardinia, in order to avoid any variability in cholesterolemia due to a different dietary response.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
decrease of LDL-cholesterol levels | 3 weeks
  42 adult volunteers (19 male and 23 female) with diagnosed mild hypercholesterolemia (total cholesterol 220-290 mg/dL), 30-60 years of age, were recruited.Individuals with a self-reported history of diabetes, inflammatory bowel disease, pancreatitis, gallbladder or biliary disease in the past 12 months, and lactose intolerance before the screening visit were excluded. Volunteers with the following characteristics were also excluded: total cholesterol ≥300 mg/dL, serum triglycerides ≥250 mg/dL or ≤ 200 mg/dL, HDL ≥70mg/dL, BMI ≥ 30, or uncontrolled hypertension at screening.

SECONDARY OUTCOMES:
endocannabinoid levels | 3 weeks
  Modification of endocannabinoid levels during intake of CLA enriched cheese.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Banni, PHD, Study Chair — Department of biomedical sciences University of Cagliari, Italy
Locations (1):
- Metabolic diseases Center AOBrotzu, Cagliari, Italy